CLINICAL TRIAL: NCT06851442
Title: A Phase Ib/II Clinical Trial to Evaluate the Efficacy and Safety of TQB3912 Tablets in Combination With Fulvestrant Injection± TQB3616 Capsules in Patients With Locally Advanced or Metastatic HR-positive and HER2-negative Breast Cancer.
Brief Title: Clinical Trial of Evaluating TQB3912 Tablets Combined With Fulvestrant Injection±TQB3616 Capsules for Locally Advanced or Metastatic Hormone Receptor(HR)-Positive and Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was closed due to business reasons. Closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3912-TQB3616-Ib/II-01
Record Dates: First submitted 2025-02-22; First posted 2025-02-28 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3912 tablets in combination with fulvestrant injection± TQB3616 capsules (Experimental): TQB3912 tablets 120 mg quaque die (QD), + fulvestrant injection 500 mg quaque 4 week(Q4W) (C1D15),28 days as a treatment cycle. Or TQB3912 tablets 120 mg quaque die(QD)+TQB3616 capsules 80 mg/120 mg QD +fulvestrant injection 500 mg quaque 4 week(Q4W) (C1D15), 28 days as a treatment cycle.
  Interventions: Drug: TQB3912 tablets in combination with fulvestrant injection± TQB3616 capsules

INTERVENTIONS:
Drug: TQB3912 tablets in combination with fulvestrant injection± TQB3616 capsules — Protein kinase B(AKT) inhibitors+Cyclin-dependent kinase 4/6(CDK4/6) Inhibitor+Estrogen receptor antagonists.

SUMMARY:
This trial was designed to evaluate the maximum tolerated dose (MTD) and phase II recommended dose (RP2D) in subjects with TQB3912 tablets combined with fulvestrant injection and TQB3616 capsules for locally advanced or metastatic HR-positive and HER2-negative breast cancer.And the effectiveness of TQB3912 tablets combined with fulvestrant injection ±TQB3616 capsules in locally advanced or metastatic HR-positive and HER2-negative breast cancer subjects was evaluated by evaluating ORR, PFS, DOR, DCR, CBR, OS, etc., and at the same time, Assess its safety and pharmacokinetic (PK) characteristics.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed an informed consent form, and had good compliance.
* Age: 18-75 years old; Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score: 0~1 point; estimated survival time exceeds 3 months.
* Women can be in the late period of menopause and before menopause/innerspring. If they are before menopause/siege period, they must continue to receive ovarian function inhibitory treatment during the research period to enter the group.
* Anthropologically confirmed HR-positive and HER2-negative breast cancer.
* Locally advanced or metastatic diseases that cannot undergo radical surgery.
* Queue 1 Previous treatment requirements: progress after endocrine therapy; Queue 2 Previous treatment requirements: progress after endocrine therapy.
* Have one or more phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA)/v-akt murine thymoma viral oncogene homolog 1 (AKT1)/phosphatase and tensin homolog deleted on chromosome ten (PTEN) gene mutations.
* At least one measurable lesion exists according to the RECIST 1.1 standard.
* Good function of the main organs
* Female subjects of childbearing age should agree that contraceptive measures (such as Buds, contraceptives or condoms) must be used during the study period and within 6 months after the study ends; the serum pregnancy test is negative within 7 days before the study enrollment. , and must be non-lactation subjects; male subjects should agree to adopt contraceptive measures within 6 months after the end of the study period.

Exclusion Criteria:

* It is known to suffer from spinal cord compression, cancerous meningitis, symptoms with brain metastasis or symptoms control for less than 4 weeks.
* Combined diseases and medical history:

  1. Have appeared within 3 years or have also suffered from other malignant tumors;
  2. Adverse reactions from previous treatments have not been restored to CTCAE 5.0 grade≤1;
  3. It affects oral and drug absorption
  4. Those who have received major surgical treatment within 4 weeks before the first medication, obvious traumatic injury or expected to undergo major surgery during the study treatment, or have long-term uncured wounds or fractures;
  5. Congenital bleeding , coagulation dysfunction disease;
  6. Arterial/deep thrombosis events occurred;
  7. Blood pressure control was not ideal;
  8. Major cardiovascular disease;
  9. Uncontrolled ≥CTCAE level 2 within 14 days before the start of study treatment
  10. A history of active tuberculosis, pulmonary fibrosis or pneumonia;
  11. a past or currently associated with interstitial lung disease/pneumonia;
  12. active viral hepatitis and poor control;
  13. treatment is required
  14. uncontrollable kidney disease;
  15. a history of immunodeficiency;
  16. a person who is prepared to undergo or has undergone genealogical bone marrow transplants or solid organ transplants;
  17. uncontrollable diabetes;
  18. a person who suffers from People with epilepsy and need treatment;
  19. People with a history of psychotropic substance abuse and cannot be abstained or have mental disorders.
* Tumor-related symptoms and treatment:

  1. If it is not controlled, the third gap effusion still needs to be repeatedly drained;
  2. There is lung cancer pharyngitis;
  3. During the study period, the tumor is very likely to invade important blood vessels and cause it Fatal severe bleeding;
  4. Use strong CYP3A4 inhibitor or strong inducer, and the drug half-life is less than 3 before the start of the study treatment;
  5. Have received anti-tumor treatment within 3 weeks before the start of the study treatment, and the washing is calculated from the end of the last treatment
  6. Within 2 weeks before the start of the study treatment, Chinese patent medicine treatment with anti-tumor indications was received in the National Medical Products Administration (NMPA) approved drug instructions.
* Research and treatment related:

  1. Used phosphatidylinositol 3 kinase (PI3K)/AKT/mammalian target of rapamycin (mTOR) inhibitors;
  2. Used fulvestrant or other selective estrogen receptor degrading agents (SERD);
  3. Used in any study drug or drug Allergic to any ingredient or excipient;
  4. a history of live attenuated vaccination within 28 days before the first medication or planned to undergo live attenuated vaccination during the study period;
  5. is receiving systemic glucocorticoid therapy or any other form of immunosuppression therapy, and Continued use within 2 weeks before the start of the study treatment
* According to the judgment of the researcher, there are situations that seriously endanger the safety of the subject or affect the subject's completion of the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 4 months after Queue 2 begins enrollment
  Phase Ib of Queue 2maximum tolerated dose (MTD, if any)
phase II recommended dose (RP2D) | 4 months after Queue 2 begins enrollment
  Phase II Queue 2: phase II recommended dose (RP2D).
Objective Remission Rate (ORR) | 8 to 16 weeks after enrollment
  Cohort 1, Phase II of Cohort 2: Objective Remission Rate (ORR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From enrollment to disease progression, an average of 14 months
  Refers to the time from the beginning of the first treatment to the first progression of the disease or death for any cause (whichever occurs first).
Duration of response (DOR) | From enrollment to disease progression, an average of 14 months
  Patient from the date of first documentation of objective remission of the tumor to the date of first documentation of objective progression of the tumor or the date of death due to any cause.
Disease control rate (DCR) | 8 to 16 weeks after enrollment
  Proportion of participants with complete response, partial response, and stable disease as rated by RECIST v1.1 criteria for best overall efficacy after enrollment of all patients.
Clinical benefit ratio (CBR) | ≥24 weeks after enrollment
  Refers to the percentage of subjects with complete remission (CR), partial remission (PR), or stable disease (SD) determined by the investigator based on RECIST 1.1 for 24 weeks.
Overall survival (OS) | From enrollment to subject death, it is expected to be evaluated until 5 years
  The time from randomization to death due to any cause.
Number of patients with adverse events (AEs) and serious adverse events (SAEs) | Within 28 days after dosing
  Assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Peak time (Tmax) | Within 24 hours after dosing
  Refers to the time after a single dose, the blood drug concentration reaches its peak.
Peak concentration (Cmax) | 30 minuets pre-dose at cycle 1 day 1, 8 and day 28. 30 minuets,1, 2, 3, 4, 6, 8, 12, 24 hours after dose at cycle 1 day 1 and day 28. Each cycle is 28 days
  Maximum plasma drug concentration.
Elimination half life (t1/2) | Within 1～7 days after dose
  The time it takes for the drug to eliminate half of the body, or the time it takes for the blood drug concentration to be reduced by half.
Area under plasma concentration-time curve (AUC0-∞) | Within 28 days after dosing
  The first dosing begins to extrapolate to an infinity plasma concentration-area under the time curve.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Fuzhou First General Hospital, Fuzhou, Fujian
  - Quanzhou First Hospital, Quanzhou, Fujian
  - Meizhou peoples Hospital, Meizhou, Guangdong
  - Guizhou Medical University Affiliated Cancer Hospital Co., Ltd, Guiyang, Guizhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Harbin Medical University Cancer, Harbin, Heilongjiang
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Yongzhou Central Hospital, Yongzhou, Hunan
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Affiliated Cancer Hospital, Ürümqi, Xinjiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Taizhou Central Hospital (Taizhou University Affiliated Hospital), Taizhou, Zhejiang